CLINICAL TRIAL: NCT06870201
Title: Dietary Iron Absorption From Lipid-Based Nutrient Supplements - A Pilot Study
Brief Title: Iron Absorption From Lipid-Based Nutrient Supplements
Status: Active, not recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other)
Responsible Party: Principal Investigator, Stephen Hennigar, Associate Professor, Pennington Biomedical Research Center
Other Study IDs: JKU/2/4/896B
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Undernutrition; Healthy
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Apparently Healthy
  Interventions: Dietary Supplement: Lipid-Based Nutrient Supplement
- Undernourished
  Interventions: Dietary Supplement: Lipid-Based Nutrient Supplement

INTERVENTIONS:
Dietary Supplement: Lipid-Based Nutrient Supplement — LNS labeled with a stable iron isotope

SUMMARY:
The overall objective of this study is to determine dietary iron absorption from lipid-based nutrient supplements (LNS) in apparently healthy and undernourished children. This case-control study will recruit apparently healthy children and children with uncomplicated undernutrition (age 1-3 years, n=15/group) from Msambweni and the surrounding rural communities in Kwale County, Kenya. At the baseline visit (day 0), participants will be provided with an LNS labeled with a stable iron isotope (57-Fe). Participants will return to the hospital 14 days later (day 14) for a blood draw. Blood collected on day 14 will be used to measure iron isotope incorporation into red blood cells. Blood collected at screening will be used to measure indicators of anemia, iron status, hepcidin, and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Children age 1-3 years on day of screening visit
* Hemoglobin 8-11 g/dL on day of screening visit
* Undernourished [length/height-for-age z-score (HAZ), weight-for-age z-score (WAZ), and/or weight-for-height/length z-score (WHZ) < -2] OR apparently healthy (HAZ, WAZ, and/or WHZ ≥ -1)

Exclusion Criteria:

* Severe acute malnutrition (WHZ < -3) with no appetite
* Serious medical condition or other chronic disease besides undernutrition (e.g., HIV+, severe pneumonia, malaria)
* Peanut allergy or other allergy that prevents consumption of the LNS
* Plans to move away from the study location during the study period

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be recruited from Msambweni and the surrounding rural communities in Kwale County, Kenya.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Dietary iron absorption | Isotope incorporation into RBCs on day 14

SECONDARY OUTCOMES:
Hemoglobin | Measured at screening
  Hemoglobin concentration
Serum ferritin | Measured at screening
  Serum ferritin concentration
Soluble transferrin receptor | Measured at screening
  Soluble transferrin receptor concentration
Transferrin saturation | Measured at screening
  Transferrin saturation percentage
Hepcidin | Measured at screening
  Hepcidin concentration
C-reactive protein | Measured at screening
  C-reactive protein concentration
Alpha-1-acid glycoprotein | Measured at screening
  Alpha-1-acid glycoprotein concentration

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hennigar, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Msambweni County Referral Hospital, Msambweni, Kenya

IPD SHARING:
Plan to Share IPD: No